CLINICAL TRIAL: NCT03256552
Title: A Randomized, Double-Blind, Chronic Dosing (7-Day), Four-Period, Four-Treatment, Placebo-Controlled, Cross-Over, Multi-Center Study to Assess the Efficacy and Safety of Three Doses of PT001 in Japanese Subjects With Moderate to Severe COPD
Brief Title: Study to Assess the Efficacy and Safety of Three Doses of PT001 in Japanese Subjects With Moderate to Severe COPD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pearl Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PT001004
Record Dates: First submitted 2017-08-17; First posted 2017-08-22 (Actual); Results first posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2017-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, chronic-dosing (7-day), four-period, four-treatment, placebo-controlled, crossover, multi-center
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- GP MDI 28.8 micrograms (Active Comparator): Glycopyrronium Metered Dose Inhaler 28.8 micrograms
  Interventions: Drug: Glycopyrronium MDI 28.8 micrograms
- GP MDI 14.4 micrograms (Active Comparator): Glycopyrronium Metered Dose Inhaler 14.4 micrograms
  Interventions: Drug: Glycopyrronium MDI 14.4 micrograms
- GP MDI 7.2 micrograms (Active Comparator): Glycopyrronium Metered Dose Inhaler 7.2 micrograms
  Interventions: Drug: Glycopyrronium MDI 7.2 micrograms
- Placebo MDI (Placebo Comparator): Placebo Inhalation Aerosol
  Interventions: Drug: Placebo MDI

INTERVENTIONS:
Drug: Glycopyrronium MDI 28.8 micrograms — Glycopyrronium MDI 28.8 micrograms
  Arms: GP MDI 28.8 micrograms
Drug: Glycopyrronium MDI 14.4 micrograms — Glycopyrronium MDI 14.4 micrograms
  Arms: GP MDI 14.4 micrograms
Drug: Glycopyrronium MDI 7.2 micrograms — Glycopyrronium MDI 7.2 micrograms
  Arms: GP MDI 7.2 micrograms
Drug: Placebo MDI — Placebo Inhalation Aerosol
  Arms: Placebo MDI

SUMMARY:
The overall objective of this study was to assess the efficacy and safety of GP MDI relative to placebo in Japanese subjects with moderate to severe COPD. Each subject received the 4 separate study treatments, scheduled as four, 7-day, treatment periods for a total treatment duration of 28 days.

DETAILED DESCRIPTION:
This was a randomized, double-blind, chronic-dosing (7-day), four-period, four-treatment, placebo-controlled, crossover, multi-center study to assess the efficacy and safety of 3 doses of GP MDI (28.8, 14.4, and 7.2 μg ex-actuator, BID) in Japanese subjects with moderate to severe COPD.

Subjects who met the entry criteria had their maintenance therapy for COPD adjusted, as specified in the protocol. To allow for an adequate washout of previous maintenance medications, subjects underwent a washout period of at least 7 days, but not greater than 28 days duration prior to returning to the clinic for Visit 2 (Randomization Visit; Day 1 of Treatment Period 1).

The 4 study treatments were GP MDI 28.8, 14.4, and 7.2 μg ex-actuator, and Placebo MDI BID. Subjects were randomly assigned to 1 of the following 4 treatment sequences (ABCD, BDAC, CADB, DCBA) in a 1:1:1:1 ratio using an Interactive Web Response System where each letter represented 1 of the 4 treatments included in the study by random assignment.

Subjects were to complete 7 days of dosing in each of the 4 Treatment Periods, with each Treatment Period separated by a washout period of 5 to 21 days.

ELIGIBILITY:
Inclusion Criteria:

* Clinical history of COPD with a moderate to severe classification
* Current and former smokers with a history of at least 10 pack-years of cigarette smoking.

-Post-bronchodilator FEV1 must be ≥30% and <80% predicted normal value-

Exclusion Criteria:

* Pregnancy
* Primary asthma diagnosis; Poorly controlled COPD defined as acute worsening of COPD that required treatment with corticosteroids or antibiotics in the 6-week interval prior to Screening or between Screening and Visit 2;
* Clinically significant abnormal ECG
* Other active pulmonary disease such as active tuberculosis, lung cancer, bronchiectasis, sarcoidosis, lung fibrosis, primary pulmonary hypertension, interstitial lung disease, and uncontrolled sleep apnea; Cancer that was not in complete remission for at least 5 years;
* Diagnosis of angle closure glaucoma
* A documented myocardial infarction within 1 year of Screening.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2015-01-28 (Actual); Primary Completion 2015-09-05 (Actual); Study Completion 2015-09-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (18):
- Japan (18):
  - Pearl Investigative Site, Fukuoka, Fukuoka
  - Pearl Investigative Site, Iizuka-shi, Fukuoka
  - Pearl Investigative Site, Mizunami-shi, Gifu
  - Pearl Investigative Site, Sapporo, Hokkaido
  - Pearl Investigative Site, Ako-shi, Hyōgo
  - Pearl Investigative Site, Himeji-shi, Hyōgo
  - Pearl Investigative Site, Kakogawa-shi, Hyōgo
  - Pearl Investigative Site, Kobe, Hyōgo
  - Pearl Investigative Site, Nishinomiya-shi, Hyōgo
  - Pearl Investigative Site, Naka-gun, Ibaraki
  - Pearl Investigative Site, Kawasaki-shi, Kanagawa
  - Pearl Investigative Site, Kyoto, Kyoto
  - Pearl Investigative Site, Kasaoka-shi, Okayama-ken
  - Pearl Investigative Site, Kishiwada-shi, Osaka
  - Pearl Investigative Site, Osaka, Osaka
  - Pearl Investigative Site, Hamamatsu, Shizuoka
  - Pearl Investigative Site, Chūōku, Tokyo-To
  - Pearl Investigative Site, Toshima-ku, Tokyo-To

REFERENCES:
- [Derived] Fukushima Y, Nakatani Y, Ide Y, Sekino H, St Rose E, Siddiqui S, Maes A, Reisner C. Randomized, double-blind, placebo-controlled trial to assess the efficacy and safety of three doses of co-suspension delivery technology glycopyrronium MDI in Japanese patients with moderate-to-severe COPD. Int J Chron Obstruct Pulmon Dis. 2018 Apr 13;13:1187-1194. doi: 10.2147/COPD.S159246. eCollection 2018. PMID 29695902

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Conducted at 20 sites in Japan from January-September 2015. Entire period of study participation per subject was a maximum of 19 weeks. Planned target enrollment of 60 subjects.
Pre-assignment Details: This was a chronic dosing (7 days), 4-period, 4-treatment, placebo-controlled, crossover study. Each subject was randomized to 1 of 4 sequences. Each sequence included the four treatment groups. By-treatment sequence tabulations of the data were not pre-specified.
Units Other Than Participants: Participants
Groups:
- Overall Study: All Subjects Randomized
Period: Overall Study
Arm/Group | Overall Study
Started | 66; 66 Participants
GP MDI 28.8 µg (Glycopyrronium Metered Dose Inhaler (MDI) 28.8 µg BID) | 61; 61 Participants
GP MDI 14.4 µg (Glycopyrronium Metered Dose Inhaler (MDI) 14.4 µg BID) | 63; 63 Participants
GP MDI 7.2 µg (Glycopyrronium Metered Dose Inhaler (MDI) 7.2 µg BID) | 62; 62 Participants
Placebo MDI (Placebo Metered Dose Inhaler BID) | 65; 65 Participants
Completed | 61; 61 Participants
Not Completed | 5; 5 Participants
Not completed — Protocol Violation | 1
Not completed — Physician Decision | 1
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: MITT Population defined as all subjects who received treatment and had post-treatment efficacy data from at least two treatment periods.
Groups:
- All Subjects: All Subjects in the MITT Population
Arm/Group | All Subjects
Number analyzed (Participants) | 62
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.5 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 59

OUTCOME MEASURES:

1. Primary Outcome: Morning Pre-dose Trough FEV1
Description: Change from Baseline in Morning Pre-dose Trough FEV1
Time Frame: Baseline, Day 8
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Groups:
- GP MDI 28.8 µg: Glycopyrronium MDI 28.8 µg
- GP MDI 14.4 µg: Glycopyrronium 14.4 µg
- GP MDI 7.2 µg: Glycopyrronium 7.2 µg
- Placebo MDI: Placebo MDI
Arm/Group | GP MDI 28.8 µg | GP MDI 14.4 µg | GP MDI 7.2 µg | Placebo MDI
Number analyzed (Participants) | 61 | 61 | 62 | 61
Liters | 0.101 [0.068 to 0.134] | 0.098 [0.066 to 0.131] | 0.077 [0.045 to 0.110] | -0.031 [-0.064 to 0.002]

2. Secondary Outcome: FEV1 AUC0-2
Description: Change from Baseline in FEV1 AUC0-2 normalized for length of follow-up. FEV1 was measured at 15 min, 30 min, 1 hour, and 2 hours post dose.
Time Frame: Day 1 and Day 8
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | GP MDI 28.8 µg | GP MDI 14.4 µg | GP MDI 7.2 µg | Placebo MDI
Number analyzed (Participants) | 61 | 61 | 62 | 62
Liters
  Day 1 | 0.176 [0.146 to 0.205] | 0.140 [0.111 to 0.170] | 0.127 [0.098 to 0.157] | 0.043 [0.014 to 0.073]
  Day 8 | 0.194 [0.157 to 0.230] | 0.199 [0.162 to 0.236] | 0.170 [0.133 to 0.206] | 0.019 [-0.018 to 0.055]

3. Secondary Outcome: Peak Change in FEV1
Description: Peak Change from Baseline in FEV1
Time Frame: Day 1 and Day 8
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | GP MDI 28.8 µg | GP MDI 14.4 µg | GP MDI 7.2 µg | Placebo MDI
Number analyzed (Participants) | 61 | 61 | 62 | 62
Liters
  Day 1 | 0.254 [0.219 to 0.289] | 0.212 [0.177 to 0.247] | 0.192 [0.157 to 0.227] | 0.104 [0.069 to 0.139]
  Day 8 | 0.260 [0.219 to 0.301] | 0.265 [0.224 to 0.306] | 0.238 [0.197 to 0.279] | 0.082 [0.041 to 0.124]

4. Secondary Outcome: FVC AUC0-2
Description: Change from Baseline in FVC AUC0-2 on Day 8 normalized for length of follow-up. FVC was measured at 15 min, 30 min, 1 hour, and 2 hours post dose.
Time Frame: Baseline, Day 8
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | GP MDI 28.8 µg | GP MDI 14.4 µg | GP MDI 7.2 µg | Placebo MDI
Number analyzed (Participants) | 61 | 61 | 62 | 61
Liters | 0.273 [0.207 to 0.339] | 0.265 [0.199 to 0.331] | 0.223 [0.157 to 0.288] | 0.047 [-0.019 to 0.113]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time the subject signed consent up to the follow-up visit 7-14 days after last dose of study drug.
Description: Safety population included all participants who received at least one dose of investigational drug and had safety data available; participants were included in safety population according to the investigational drug received
Arm/Group | GP MDI 28.8 µg | GP MDI 14.4 µg | GP MDI 7.2 µg | Placebo MDI
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/63 | 0/62 | 1/65
Other Adverse Events (participants affected / at risk) | 2/61 | 2/63 | 1/62 | 1/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GP MDI 28.8 µg (N=61) | GP MDI 14.4 µg (N=63) | GP MDI 7.2 µg (N=62) | Placebo MDI (N=65)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GP MDI 28.8 µg (N=61) | GP MDI 14.4 µg (N=63) | GP MDI 7.2 µg (N=62) | Placebo MDI (N=65)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Drafts of any and all publications or presentations of this study must be submitted at least 30 days prior to submission for publication or presentation to Pearl Therapeutics for review, approval, and to ensure consistency. Pearl Therapeutics has the right to request appropriate modification to correct facts and to represent its opinions, or the opinions of the publication committee, if these differ with the proposed publication.